CLINICAL TRIAL: NCT04802395
Title: Real World Evidence Clinical Utility Study of KidneyIntelX in Patients With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: Real World Evidence Clinical Utility Study of KidneyIntelX
Status: Recruiting | Type: Observational
Sponsor: Renalytix AI, Inc. (Industry)
Collaborators: Mount Sinai Hospital, New York (Other)
Responsible Party: Sponsor
Other Study IDs: RAI 19-1004
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases; Diabetic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: KidneyIntelX — KidneyIntelX is an in-vitro diagnostic that enables accurate risk prediction of progressive decline in kidney function in patients with type 2 diabetes and existing CKD at stages 1-3 (eGFR of 30 to 59 ml/min/1.73m2, or eGFR ≥ 60 ml/min/1.73m2 and uACR ≥ 30 mg/g).

SUMMARY:
The purpose of this study is to assess the impact of the KidneyIntelX assay utilized as part of the current standard of care on the management of patients seen in the primary care physician's office at Mount Sinai.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Type 2 diabetes and concurrent chronic (diabetic) kidney disease (G3a-G3b or G1-G2, A2-A3) per KDIGO CKD staging.

Exclusion Criteria:

* Patents without the appropriate characteristics as identified in the KidneyIntelX intended use population.
* Patients with eGFR <30 or ≥ 60 ml/min/1.73m2 without albuminuria.
* Patients with ESRD or on renal recovery treatments at time of enrollment.
* Patients who are pregnant at the time of enrollment.
* Patients who are currently hospitalized.
* Patients without minimum 6 month pre-baseline KidneyIntelX medical history.
* Patients who are currently on Enbrel.

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes and existing chronic kidney disease stages 1-3.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Referrals | 6 Months
  Proportion (target: 20%) of patients referred to a dietician, diabetologist, or nephrologist.
Statins and or ACEi/ARB | 6 Months
  Proportion (target: 20% increase) of patients treated with statins and or angiotensin-converting-enzyme inhibitors and angiotensin II receptor blockers.
HbA1c | 6 Months
  Proportion (target: 20% increase) of patients to receive information and or advice on their individualized target of HbA1c.
SGLT2/ GLP1 | 6 Months
  Proportion (target: 20% increase) of patients treated with SGLT2 inhibitors or GLP1 agonists.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided